CLINICAL TRIAL: NCT06734000
Title: Cohorte COSCINUS - Biocollection COhort in Spinal Cord Injury - Nantes Follow-Up Standardization
Brief Title: Cohorte COSCINUS - Biocollection
Acronym: COSCINUS
Status: Recruiting | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC24_0413; 2024-A01711-46 (Other: ANSM)
Record Dates: First submitted 2024-10-09; First posted 2024-12-13 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2024-12

CONDITIONS: Spinal Cord Injury
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples Without DNA — Blood, urine and stool
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Individuals with spinal cord injury: Collection of blood, urine and feces during the 5 years after the lesion.

SUMMARY:
COSCINUS is a standardized framework for evaluating temporal trends in SCI causes, SCI characteristics, and demographic patterns. It allows a precise estimation of medical complications' incidence, their evolution over time, as well risk factors influencing these complications, including management modalities. Moreover, COSCINUS provides a high-quality research platform, including clinical, epidemiological, biostatistical, and IT expertise, thereby promoting fundamental research in spinal cord injury and related autonomic dysfunctions. As a national epidemiological tool, COSCINUS offers unique analytical perspectives, promising significant contributions to the understanding and management of spinal cord injuries.

DETAILED DESCRIPTION:
The Neurological Physical and Rehabilitation Medicine (NPRM) Department at Nantes University Hospital, referral centre for SCI patients, has been working since 2015 on the creation of a comprehensive database. This database systematically collects a wide range of data, including socio-demographic, clinical, health status, activity and participation data for SCI patients.

Paired with this database is a longitudinal biocollection that preserves blood, urinary, and feces samples enabling analyses of the microbiome, biomarkers as metabolic, inflammatory, immune, and injury severity biomarkers.

The COSCINUS cohort and its biocollection, created through a multidisciplinary approach, are longitudinally structured. They entail meticulous and continuous recording of standardized data and specific sample collection across various phases of spinal cord injury management, from the acute phase through long-term follow-up.

Data and samples are collected prospectively at specific time points:

Acute phase, admission to PRM department, 6 months post-injury, discharge and during scheduled follow-up consultations (1 / 2 / 3 years post-injury…) with additional collection in case of complications

ELIGIBILITY:
Inclusion Criteria:

* All individuals with spinal cord injury admitted to the neurological PRM department of the Nantes University Hospital at the initial phase of development of the paraplegia or tetraplegia could participate, regardless the clinical neurological status.

Exclusion Criteria:

* Patients not covered by social security.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All individuals with spinal cord injury admitted to the neurological PRM department of the Nantes University Hospital at the initial phase of development of the paraplegia or tetraplegia could participate, regardless the clinical neurological status.
Sampling Method: Non-Probability Sample
Enrollment: 105 (Estimated)
Dates: Start 2024-12-13 (Actual); Primary Completion 2032-10-10 (Estimated); Study Completion 2032-10-10 (Estimated)

PRIMARY OUTCOMES:
Dosage of urinary polyunsaturated fatty acid derivatives | 5 years
  Urinary biocollection: correlate the evolution of urinary PUFAs and urinary microbiota with the type of neurovessel, mictional mode, complications, notably infectious, and response to treatment of neurogenic detrusor overactivity (anticholinergic, intra-detrusor botulinum toxin) through data sets: lower urinary tract function, lower urinary tract urodynamics, urinary infections, urinary tree imaging and bladder toxin injection follow-up.
Analysis of fecal polyunsaturated fatty acid derivatives | 5 years
  Fecal biocollection: correlate evolution of fecal microbiota and evolution of polyunsaturated fatty acids in stool with severity of digestive disorders using the International Spinal Cord Injury and Bowel Function data set including the Neurogenic Bowel Dysfunction score.
Analysis of the blood biomarker's evolution in individuals with a spinal cord injury from the injury | 5 years
  Blood biocollection: correlating bone resorption markers with fracture datasets and immunological status with Autonomic nervous system and antibiotic therapy datasets
Analysis of the biomarker's evolution in individuals with a spinal cord injury from the injury | 5 years
  This longitudinal analysis will correlate the evolution of biomarkers reflecting neurological and systemic impairments with their severity and treatment response, including the patient's neurological status (neurological level of the lesion, completeness, and evolution assessed by ISNCSCI)

CONTACTS AND LOCATIONS:
Locations (1):
- Nantes University Hospital, Nantes, Loire-Atlantique, France

IPD SHARING:
Plan to Share IPD: Undecided